CLINICAL TRIAL: NCT02939716
Title: A Pilot Study to Assess the Effect of Lettuce on Intestinal Water Content Through Magnetic Resonance Imaging of the Small Bowel: LETIS
Brief Title: Assessing the Effect of Lettuce on Intestinal Water Content Through Magnetic Resonance Imaging of the Small Bowel
Acronym: LETIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Responsible Party: Principal Investigator, Robin Spiller, Professor of Gastroenterology, University of Nottingham
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: C12072016 MRI
Record Dates: First submitted 2016-10-13; First posted 2016-10-20 (Estimated); Results first posted 2020-07-31 (Actual); Last update posted 2020-07-31 (Actual); Status verified 2020-07

CONDITIONS: Asymptomatic Conditions
Keywords: small bowel; bloating; flow
MeSH Terms: conditions — Asymptomatic Diseases | interventions — rhubarb peony decoction; Bread

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Rhubarb (Active Comparator): 300g frozen rhubarb, microwaved; served with 65g lactose free cream and saccharine sweetener
  Interventions: Other: Rhubarb
- Bread (Active Comparator): 2 slices of white bread, 40g each; served with 10g butter
  Interventions: Other: Bread
- Lettuce (Experimental): 300g lettuce; served with 30g mayonnaise
  Interventions: Other: Lettuce

INTERVENTIONS:
Other: Rhubarb — 300gm rhubarb
  Arms: Rhubarb
Other: Bread — 2 slices bread
  Arms: Bread
Other: Lettuce — 300g lettuce
  Arms: Lettuce

SUMMARY:
When patients have bowel surgery they are sometimes left with a stoma, where the small bowel exits onto the wall of the abdomen, not into the colon. Certain foods have been shown to increase the amount of water lost through a stoma. This can lead to dehydration. Such patients are encouraged to avoid such foods but knowing which ones to avoid relies partly on trial and error.

In a survey 1 in 3 patients said that rhubarb increased stoma output. Rhubarb is known to contain chemicals that can stimulate the bowel. 1 in 6 patients also reported the same effect with lettuce which has not previously been shown to have such an effect. Latex found in lettuce leaves may stimulate the bowel to produce more fluid, explaining this effect.

In Nottingham the investigators have developed techniques that use Magnetic Resonance Imaging (MRI) to measure water in the small bowel. They want to use these techniques to explore whether eating lettuce increase small bowel water content. They will compare lettuce to rhubarb and to bread, which they know reduces small bowel water. They will see if they can detect any relationship between water in the bowel and feelings of bloating.

DETAILED DESCRIPTION:
Background:

In recent years fermentable oligo-, di-, mono-saccharides and polyols, have been proposed to exacerbate symptoms of irritable bowel syndrome (IBS) such as abdominal discomfort and bloating. This phenomenon has also been observed in patients with an ileostomy, where certain foods have been associated with increased fluid output from the stoma. This is in accordance with past work surveying ileostomy patients on foods that altered stoma function. However, there may be other factors that drive fluid output from a stoma. Rhubarb, a food listed by 1 in 3 patients as exacerbating watery diarrhoea, also contains anthraquinones that have laxative effects, such as in senna.

A food less commonly associated with laxative effects is lettuce but 1 in 6 patients reported that eating lettuce led to an increase in watery stoma output. Certain lettuce varieties exude a milk-like latex material when cut, giving rise to the latin name Lactuca sativa. While the methylcellulose is insoluble and would not be expected to hold water in the lumen of the small bowel, latex could be expected to stimulate intestinal secretion. This may contribute to post-prandial sensations of bloating by a different mechanism to the osmotic effects and colonic fermentation seen with poorly absorbed but fermentable carbohydrates..

The Nottingham GI MRI group has been at the forefront of elucidating the effects of poorly digested carbohydrates on gastrointestinal physiology. the investigators have published techniques to measure free water in the small bowel and assessment of viscosity in the colon using MR relaxometry. This includes the demonstration that fructose ingestion on its own leads to increased free water in the small bowel compared to co-ingestion with glucose - see panel. The investigators wish to apply these techniques to compare the effect of different foods: white bread, lettuce and rhubarb. The investigators have previously shown that bread led to a reduction in small bowel water and so can active as a negative control. Rhubarb should serve as a positive control.

Aims: The purpose of the study is gather pilot data on the effect of different foods on intestinal physiology.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 or older
* Able to give informed consent

Exclusion Criteria:

* Pregnancy declared by candidate
* History declared by the candidate of pre-existing gastrointestinal disorder that may affect bowel function
* A positive diagnosis of irritable bowel syndrome based on the Rome III criteria questionnaire
* Reported history of previous resection of the oesophagus, stomach or intestine (excluding appendix)
* Intestinal stoma
* Any medical condition making participation potentially compromising participation in the study e.g. diabetes mellitus, respiratory disease limiting ability to lie in the scanner, known allergy to one of the food products
* Contraindications for MRI scanning i.e. metallic implants, pacemakers, history of metallic foreign body in eye(s) and penetrating eye injury
* Will not agree to dietary restrictions required in 24 hours before each study day
* Unable to stop drugs known to alter GI motility including mebeverine, opiates, monoamine oxidase inhibitors, phenothiazines, benzodiazepines, calcium channel antagonists for the duration of the study (Selective serotonin reuptake inhibitors and low dose tricyclic antidepressants will be recorded but will not be an exclusion criteria)
* Inability to lie flat or exceed scanner limits of weight <120kg
* Poor understanding of English language
* Participation in night shift work the week prior to the study day. Night work is defined as working between midnight and 6.00 in the morning
* Participation in any medical trials for the past 3 months
* Anyone who in the opinion of the investigator is unlikely to be able to comply with the protocol e.g. cognitive dysfunction, chaotic lifestyle related to substance abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2016-10; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robin Spiller, Principal Investigator — University of Nottingham
Locations (2):
- United Kingdom (2):
  - Sir Peter Mansfield Imaging Centre, Nottingham
  - Nottingham Digestive Diseases Centre, Nottingham

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 15 included in final analysis as scanner failure caused loss of data for 3 subjects
Groups:
- Healthy Volunteers. Bread Then Lettuce Then Rhubarb: Healthy volunteers free from GI disease. Randomised to order Bread then Lettuce then Rhubarb
- Healthy Volunteers. Bread Then Rhubarb Then Lettuce: Healthy volunteers free from GI disease. Randomised to order Bread then Rhubarb then Lettuce
- Healthy Volunteers. Lettuce Then Rhubarb Then Bread: Healthy volunteers free from GI disease. Randomised to order Lettuce then Rhubarb then Bread
- Healthy Volunteers. Lettuce Then Bread Then Rhubarb: Healthy volunteers free from GI disease. Randomised to order Lettuce then Bread then Rhubarb
- Healthy Volunteers. Rhubarb Then Bread Then Lettuce: Healthy volunteers free from GI disease. Randomised to order Rhubarb then Bread then Lettuce
- Healthy Volunteers. Rhubarb Then Lettuce Then Bread: Healthy volunteers free from GI disease. Randomised to order Rhubarb then Lettuce then Bread
Period: Overall Study
Arm/Group | Healthy Volunteers. Bread Then Lettuce Then Rhubarb | Healthy Volunteers. Bread Then Rhubarb Then Lettuce | Healthy Volunteers. Lettuce Then Rhubarb Then Bread | Healthy Volunteers. Lettuce Then Bread Then Rhubarb | Healthy Volunteers. Rhubarb Then Bread Then Lettuce | Healthy Volunteers. Rhubarb Then Lettuce Then Bread
Started | 3 | 3 | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 2 | 2 | 2
Not Completed | 0 | 0 | 0 | 1 | 1 | 1
Not completed — scanner failure | 0 | 0 | 0 | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Healthy Volunteers: Healthy volunteer group who participated
Arm/Group | Healthy Volunteers
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 15

OUTCOME MEASURES:

1. Primary Outcome: Small Bowel Water Content Measured by MRI
Description: Area under the curve of postprandial change from fasting small bowel water, 0-3 hours, measured by MRI, in mL*min
Time Frame: 0-3 hours
Population: 15 healthy volunteers free from GI disorders.
Measure: Mean (Standard Error); unit: mL*min
Groups:
- Healthy Volunteers. Bread Arm.: Bread Arm.
- Healthy Volunteers. Lettuce Arm: Lettuce Arm
- Healthy Volunteers. Rhubarb Arm: Rhubarb Arm
Arm/Group | Healthy Volunteers. Bread Arm. | Healthy Volunteers. Lettuce Arm | Healthy Volunteers. Rhubarb Arm
Number analyzed (Participants) | 15 | 15 | 15
mL*min | -5662 (1209) | 3194 (1574) | 10586 (1629)

2. Secondary Outcome: Ascending Colon Water Content
Description: Area under the curve of postprandial change from fasting ascending colon water, 0-3 hours, measured by MRI, in mL*min
Time Frame: 0-3 hours
Population: Healthy Volunteers
Measure: Mean (Standard Error); unit: mL*min
Groups:
- Bread: Bread Arm
- Lettuce: Lettuce Arm
- Rhubarb: Rhubarb Arm
Arm/Group | Bread | Lettuce | Rhubarb
Number analyzed (Participants) | 15 | 15 | 15
mL*min | 78 (43) | 409 (231) | 291 (89)

3. Secondary Outcome: Relaxation Time in Ascending Colon
Description: Area under the curve of postprandial change from fasting small bowel water, 0-3 hours, measured by MRI in milliseconds.min
Time Frame: 0-3 hours
Population: Healthy volunteers free from GI disorders
Measure: Mean (Standard Error); unit: ms*min
Arm/Group | Bread | Lettuce | Rhubarb
Number analyzed (Participants) | 15 | 15 | 15
ms*min | 15188 (6717) | 18990 (7884) | 35744 (9013)

4. Secondary Outcome: Bloating VAS Score
Description: Area under the curve of postprandial change from fasting bloating score, 0-180 min, measured by a 100 point visual analogue scale (VAS), where 0 is no symptom and 100 is worst symptom. Measured every 30 mins.
Time Frame: 0-180 min
Population: Healthy volunteers
Measure: Mean (Standard Error); unit: VAS Score*Min
Arm/Group | Bread | Lettuce | Rhubarb
Number analyzed (Participants) | 15 | 15 | 15
VAS Score*Min | 4196 (637) | 7071 (905) | 5113 (927)

5. Secondary Outcome: Satiety VAS Score
Description: Area under the curve of postprandial change from fasting satiety score, 0-180 min, measured by a 100 point visual analogue scale (VAS), where 0 is no symptom and 100 is worst symptom. Measured every 30 mins.
Time Frame: 0-180 mins
Population: Healthy volunteers free from GI disorders
Measure: Mean (Standard Error); unit: VAS Score*Mins
Arm/Group | Bread | Lettuce | Rhubarb
Number analyzed (Participants) | 15 | 15 | 15
VAS Score*Mins | 7943 (783) | 9498 (941) | 7904 (835)

ADVERSE EVENTS:
Time Frame: From initial participant recruitment visit to last participant visit. This covered 4 months from Sept 2016- January 2017. There was no follow up period.
Groups:
- Healthy Volunteers. Bread Then Lettuce Then Rhubarb: Healthy Volunteers. Treatment order Bread Then Lettuce Then Rhubarb
- Healthy Volunteers. Bread Then Rhubarb Then Lettuce: Healthy Volunteers. Treatment order Bread Then Rhubarb Then Lettuce
- Healthy Volunteers. Lettuce Then Rhubarb Then Bread: Healthy Volunteers. Treatment order Lettuce Then Rhubarb Then Bread
- Healthy Volunteers. Lettuce Then Bread Then Rhubarb: Healthy Volunteers. Treatment order Lettuce Then Bread Then Rhubarb
- Healthy Volunteers. Rhubarb Then Bread Then Lettuce: Healthy Volunteers. Treatment order Rhubarb Then Bread Then Lettuce
- Healthy Volunteers. Rhubarb Then Lettuce Then Bread: Healthy Volunteers. Treatment order Rhubarb Then Lettuce Then Bread
Arm/Group | Healthy Volunteers. Bread Then Lettuce Then Rhubarb | Healthy Volunteers. Bread Then Rhubarb Then Lettuce | Healthy Volunteers. Lettuce Then Rhubarb Then Bread | Healthy Volunteers. Lettuce Then Bread Then Rhubarb | Healthy Volunteers. Rhubarb Then Bread Then Lettuce | Healthy Volunteers. Rhubarb Then Lettuce Then Bread
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/3 | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/3 | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/3 | 0/3 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-16): https://cdn.clinicaltrials.gov/large-docs/16/NCT02939716/Prot_SAP_000.pdf